CLINICAL TRIAL: NCT02055937
Title: Immediate Implant Breast Reconstruction for Patients With Mastectomy Ans Post opérative Chest Wall Radiotherapy
Brief Title: Immediate Implant Breast Reconstruction
Acronym: ISIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: autorities vorbidden this dispositif in other trial
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VA2012/37; 2012-A01369-34 (Registry Identifier: RCB)
Record Dates: First submitted 2013-10-09; First posted 2014-02-05 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
Keywords: mastectomy, reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- immediate implant breast reconstruction (Experimental): immediate implant breast reconstruction
  Interventions: Procedure: immediate implant breast reconstruction

INTERVENTIONS:
Procedure: immediate implant breast reconstruction — Eligible patients will undergo radical mastectomy with axillary lymph nodes sampling followed by immediate and single-stage breast reconstruction using the acellular dermal matrix Strattice™

SUMMARY:
The purpose of this study is to study the impact of the immediate implant breast reconstruction for patients with mastectomy and postoperative chest wall radiotherapy

DETAILED DESCRIPTION:
non applicable

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast carcinoma
* Patients planned for mastectomy with immediate single stage breast reconstruction using an acellular dermal matrix (Strattice™, LifeCell Corporation)
* Patients planned to receive postoperative chest wall irradiation
* Age ≥ 18 years old
* WHO performance status 0-1
* Affiliation to a social security system
* Informed consent signed prior any study specific procedures

Exclusion Criteria:

* Inflammatory breast cancer
* Tumors with extensive involvement of the skin
* Use of tissue expander
* Indication of postoperative chemotherapy
* Patients planned for bilateral mastectomy
* History of previously treated ipsilateral breast carcinoma
* Usual contraindications for ADM
* Medical debility precluding surgical treatment
* Psychological, social, geographical disorders or any other condition that would preclude study compliance (treatment modalities and study follow-up).
* Pregnancy or breast feeding
* Inability to attend or comply with interventions or follow-up scheduling, disability or difficulty preventing a proper understanding of trial instructions
* Legal inability or restricted legal ability

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Success is defined as a complete therapeutic sequence (surgery + RT) without any significant complication at 6 months. | confirm the feasibility of the therapeutic sequence at 6 months
  Success is defined as a complete therapeutic sequence (surgery + RT) without any significant complication at 6 months.
  Significant complication is defined as:
  * Any event delaying RT (delay surgery/RT > 3 months)
  * Any event preventing patients from receiving radiotherapy within 6 months after surgery

SECONDARY OUTCOMES:
The rate of Baker | up to 36 months after surgery
  The rate of Baker grades 3/4 capsular contracture

OTHER OUTCOMES:
Cosmetic results | up to 36 months after surgery
  Cosmetic results: assessed by both the surgeon and patient (patient satisfaction will be evaluated using a self-questionnaire). Photographs of the breast will be taken at different times (Pre / per / postoperative) and the picture analysis will be reviewed by an independent committee.
Functional results | up to 36 months after surgery
  Functional results: patient satisfaction will be evaluated using a self-questionnaire
The rate of patients requiring breast implant removal | up to 36 months after surgery
  The rate of patients requiring breast implant removal
Study of tolerance | up to 36 months after surgery
  Study of the indesirable effect of the radiotherapy on the implant

CONTACTS AND LOCATIONS:
Locations (1):
- Institut régional du Cancer - Montpellier - Val d'Aurelle, Montpellier, France

REFERENCES:
- [Background] Christian CK, Niland J, Edge SB, Ottesen RA, Hughes ME, Theriault R, Wilson J, Hergrueter CA, Weeks JC. A multi-institutional analysis of the socioeconomic determinants of breast reconstruction: a study of the National Comprehensive Cancer Network. Ann Surg. 2006 Feb;243(2):241-9. doi: 10.1097/01.sla.0000197738.63512.23. PMID 16432358
- [Background] Lambert K, Mokbel K. Does post-mastectomy radiotherapy represent a contraindication to skin-sparing mastectomy and immediate reconstruction: an update. Surg Oncol. 2012 Jun;21(2):e67-74. doi: 10.1016/j.suronc.2011.12.007. Epub 2012 Jan 30. PMID 22296996